CLINICAL TRIAL: NCT00121875
Title: Growth Hormone and Insulin Resistance in Girls With Turner Syndrome or Idiopathic Short Stature
Brief Title: Study to Identify Markers of Insulin Resistance During Growth Hormone Treatment for Short Stature
Status: Terminated | Type: Observational
Why Stopped: Enrollment was too low.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Lynne L. Levitsky, M.D., Massachusetts General Hospital
Other Study IDs: 2004P-002800; L3452n
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Turner Syndrome; Idiopathic Short Stature
Keywords: short stature; insulin resistance; body composition; Turner syndrome; intramyocellular lipid; glucose tolerance
MeSH Terms: conditions — Turner Syndrome; Dwarfism; Insulin Resistance | interventions — Human Growth Hormone; DNA, Ribosomal; Growth Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Turner syndrome: Girls, aged 7-14, with short stature due to Turner syndrome and eligible for growth hormone therapy
  Interventions: Drug: somatropin (rDNA)
- Control / idiopathic short stature: Girls, aged 7-14, with idiopathic short stature and eligible for growth hormone therapy
  Interventions: Drug: somatropin (rDNA)

INTERVENTIONS:
Drug: somatropin (rDNA) — Form/Strength: 10 mg aqueous suspension; 5 mg/ml
  Dosage/Frequency: 0.35 mg/kg/week, daily divided doses
  Duration: 6 months with 3-month washout period
  Other Names: recombinant human growth hormone, Nutropin-AQ

SUMMARY:
Growth hormone treatment improves body fat distribution but also causes insulin resistance. Scientists have recently linked insulin resistance with special stores of fat in the muscles, which can be measured by magnetic resonance imaging (MRI). The researchers hypothesize that growth hormone will paradoxically reverse the linkage between muscle fat stores and insulin resistance. To assess this association and to investigate the cause(s), the researchers will measure muscle fat stores during growth hormone treatment. Other parameters linked to insulin resistance (glucose tolerance, blood markers, and body composition) will also be assessed. This study may lead to improved strategies for monitoring growth hormone therapy.

DETAILED DESCRIPTION:
Growth hormone (GH) treatment can cause insulin resistance (IR) despite its overall favorable influence on body fat composition. IR is associated with special stores of fat in the muscle (intramyocellular lipid or IMCL), which can be measured by MRI. The researchers hypothesize that changes in IR during GH treatment will be associated with a predictable, but possibly contradictory, change in muscle fat stores. Girls receiving GH for short stature, due to Turner syndrome or idiopathic short stature (ISS), will be studied both during and without GH treatment to assess the impact of GH treatment on muscle fat stores.

Hypothesis: Girls with Turner syndrome will have increased IMCL, corresponding to their insulin resistance, when compared to girls with ISS. GH treatment may paradoxically reverse this association in girls with Turner syndrome.

Objectives: The objectives are to assess changes in IMCL during GH therapy and to increase the researchers' knowledge of GH action.

Study Design: Prepubertal girls receiving GH therapy for short stature due to Turner syndrome or ISS will be recruited to participate in a crossover study. Subjects will be studied twice: first during GH treatment and at baseline, following washout without GH for 3 months. GH treatment for up to 6 months will be provided for eligible girls not currently receiving GH. Assessments include:

* IMCL (soleus and tibialis anterior) measured non-invasively by proton magnetic resonance spectroscopy (1H-MRS)
* Body composition measured by DEXA and morphometry
* Whole body insulin sensitivity assessed by oral glucose tolerance
* Levels of plasma lipids and hormones

Endpoints: The primary endpoint is to define the effect of GH on IMCL content in girls with Turner syndrome versus girls with ISS. The secondary endpoint is to examine how GH affects IMCL content by identifying correlative changes in plasma hormones and metabolites.

Significance: This study is intended to find improved strategies for monitoring GH therapy. In addition, IMCL is anticipated to be a valuable probe for understanding GH effects on glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Girls, with Turner syndrome or ISS; height standard deviation score (SDS) ≤ -2
* Bone age ≤ 12 years
* Normal birthweight
* Body mass index (BMI) = 10th-90th percentile
* Normal childhood activity; no physical or other limitations
* Normal, balanced diet (20-40% calories from fat)

Exclusion Criteria:

* Puberty (beyond Tanner Stage 1)
* Diabetes in subject or first degree relative
* Sex steroid therapy
* Chronic conditions requiring medication (treatment for hypothyroidism is permissible)
* Significant systemic disease (pulmonary, cardiac, renal, or other)
* Non-removable metal

Ages: 7 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Girls, age 7-14 years, with short stature due to Turner syndrome or with idiopathic short stature
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2005-06; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to compare the effect of GH on IMCL content in the two subject groups (Turner syndrome vs. ISS) | 3 months

SECONDARY OUTCOMES:
to assess the relationship of IMCL to IR-associated plasma markers in each groups | 3 months
to assess the relationship of IMCL to the effect of GH therapy in each groups | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynne L Levitsky, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States